CLINICAL TRIAL: NCT04144894
Title: The Biosonographic Index - A Novel Index for the Early Detection of Acute Kidney Injury After Vascular Surgery - an Exploratory Study.
Brief Title: The Biosonographic Index
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Ahmed Zaky, Principal Investigator, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-300003010; UAB (Other: Anesthesiology)
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Healthy Controls (Other)
  Interventions: Diagnostic Test: Shear Wave Elastography
- Vascular Surgery Subjects (Other)
  Interventions: Diagnostic Test: Shear Wave Elastography

INTERVENTIONS:
Diagnostic Test: Shear Wave Elastography — Advanced ultrasound technique

SUMMARY:
In this exploratory study we explore the use of Shear Wave Elastography to differentiate between Acute Kidney Injury after vascular surgery and among the healthy population.

ELIGIBILITY:
Inclusion Criteria:

* No history of diabetes or hypertension
* Estimated Glomerular Filtration Rate > 60 ml/min/m^2
* Structurally normal kidney on renal ultrasound
* BMI < 27 kg/m^2

Exclusion Criteria:

* Prisoners directly admitted from a correctional facility
* Children < 19 years or under 50 kg body weight if age is unknown
* Patients with end stage renal disease or preexisting glomerular filtration rate less than or equal to 30 mL/min/1.73 m^2 or need for dialysis
* Patients with end stage heart disease on the cardiac transplant list
* Patients undergoing procedures without vascular surgery
* All transplant patients
* Patients on ventricular assist devices
* Patients undergoing emergency procedures
* Patients with body mass index > 27kg/m^2
* Any condition that would impede visualization of the kidneys by ultrasound

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-12-02 (Estimated)

PRIMARY OUTCOMES:
Diagnostic factor of Shear Wave Elastography | From the time of Informed Consent being given to 96 hours after consent being given
  Shear wave Elastography-derived Young's Elastic Modulus factor differentiating patients with Acute Kidney Injury post vascular surgery from healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Zaky, MD, MPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zaky A, Beck AW, Bae S, Sturdivant A, Liwo A, Zdenek N, McAnally N, Ahmad S, Meers B, Robbin M, Pittet JF, Tolwani A, Berkowitz D. The bio-sonographic index. A novel modality for early detection of acute kidney injury after complex vascular surgery. A protocol for an exploratory prospective study. PLoS One. 2020 Nov 17;15(11):e0241782. doi: 10.1371/journal.pone.0241782. eCollection 2020. PMID 33201924